CLINICAL TRIAL: NCT05067751
Title: Evaluating the Effectiveness of Asymmetrical Directionality With Bimodal Systems.
Brief Title: Asymmetrical Directionality With Bimodal Systems.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: GN Hearing A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: Parker
Record Dates: First submitted 2021-09-21; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: hearing aid with directionality — Hearing directionality allows users the ability to focus on voices and other signals of interest, reducing background noises that are unimportant.

SUMMARY:
Research supports that bimodal stimulation includes improvements in auditory performance and daily living over using a cochlear implant (CI) or hearing aid (HA) alone. Although bimodal users continue to achieve high levels of satisfaction, speech perception in noise continues to be highly problematic. The aim of this field study is to identify which directionality schemes in a bimodal solution are preferred by users using an ecological momentary assessment tool.

DETAILED DESCRIPTION:
The primary purpose of this research trial is to evaluate asymmetrical directionality in bimodal users for hearing speech in noise in the sound field and in daily life using an EMA tool. The aim is to collect information regarding hearing for speech in background noise as well as end-user insights, testimonials, and communication content.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the inclusion criteria described below to be eligible for this clinical investigation.

1. Adults who are English speaking and aged 18 years and older.
2. Individuals with a mild sloping to severe/profound hearing loss in the hearing aided ear.
3. New and experienced bimodal users (cochlear implant + hearing aid).
4. Experienced Nucleus 7 or Kanso 2 cochlear implant users with minimum experience using electrical hearing for 6 months.
5. Individuals able to complete test measures as outlined in the informed consent and protocol.
6. Individuals with access to a Smart Phone/device that is either iOS 7.0 or Android 4.0 and later who are willing to utilize their personal Smart Phone/device for participation in the trial.
7. Individuals willing to use their personal email account for participation in the trial.

   -

Exclusion Criteria:

Subjects who meet any of the exclusion criteria described below will not be eligible for this clinical investigation.

1. Individuals using sound processors in the Hybrid mode.
2. Bilateral cochlear implant users.
3. Unable or unwilling to comply with the requirements of the study as determined by the Investigator.
4. Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
5. Currently participating, or participated within the last 30 days, in another interventional clinical investigation/trial involving an investigational device.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects, male/female with diagnosed hearing loss that have been treated with Cochlear implants in one ear.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-10-06 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Hearing loss assessed by the SSQ 12 hearing related questionnaire | 2 weeks
  Speech Spatial and Qualities of hearing questionnaire is designed to measure of range of hearing disabilities across several domains. Specific attention is given to hearing speech in a host of competing contexts, and to the directional, distance and movement components of spatial hearing.

SECONDARY OUTCOMES:
Hearing loss assessed by the AZ Bio sentence test in the presence of noise | 2 weeks
  AZ Bio sentence in noise test comprised of 15 lists of 20 sentences each and is a measure of speech perception ability by individuals that mimics real life conditions with the presence of background noise.

OTHER OUTCOMES:
Hearing loss will be assessed by using ecological momentary assessments to get a repeated sampling of their behaviors and experiences in real time. | 1 week
  Ecological momentary assessment will act as a digital diary, in real time, to understand subject's real life behaviors in their momentary environments.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Quilter, Principal Investigator — GN Hearing

IPD SHARING:
Plan to Share IPD: No